CLINICAL TRIAL: NCT00908661
Title: Study of the Effectiveness of a Lightweight Mesh (Polypropylene and Poliglecaprone 25 and Oxidized Cellulose) in the Prevention of Parastomal Hernia in Patients Requiring a Permanent Ostomy. Laparoscopic Approach
Brief Title: Effectiveness of a Lightweight Mesh in the Laparoscopic Prevention of Parastomal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: MANUEL LOPEZ-CANO, MD,PhD, Hospital Universitari Vall d'Hebron. Department of Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PR(AG)116/2006
Record Dates: First submitted 2009-05-25; First posted 2009-05-27 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2011-03

CONDITIONS: Parastomal Hernia
Keywords: Parastomal, hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylactic mesh (Active Comparator): All patients will have a permanent ostomy and a randomisation with prophylactic mesh
  Interventions: Device: Lightweight polipropilene and poliglecaprone 25 and oxidized cellulose mesh
- without prophylactic mesh (No Intervention): All patients will have a permanent ostomy and a randomisation without prophylactic mesh

INTERVENTIONS:
Device: Lightweight polipropilene and poliglecaprone 25 and oxidized cellulose mesh — Lightweight polipropilene and poliglecaprone 25 and oxidized cellulose mesh
  Other Names: PROCEED mesh
  Arms: Prophylactic mesh

SUMMARY:
The purpose of this study is to determine if a mesh is effective in the prevention of a parastomal hernia when a permanent ostomy is performed through a laparoscopic approach.

DETAILED DESCRIPTION:
Parastomal hernia (PH) is a very common complication after abdominal surgery that requires a permanent ostomy. This type of surgery is usually associated with processes that fall within the scope of Coloproctology.PH is difficult to deal with high rates of recurrence after surgical repair.This type of hernia remains a problem of first order, generating a significant consumption of health and economic resources and determining an impaired quality of life of these patients.Laparoscopic surgery is increasingly used in colorectal surgery.

Also with this type of approach is present the problem of prevention of PH. The use of a mesh in the repair of hernias is not discussed since the placement of a prosthesis significantly reduces the recurrence rate. There are now many types of prosthetic meshes available. A low weight mesh composed of large pores (about 5mm) with a high proportion of absorbable material and a layer of oxidized regenerated cellulose which is placed in the vicinity of the bowel is available on the market (PROCEED ®, Ethicon). The introduction of this low-weight mesh provides a good opportunity to prevent the development of an PH when we use a laparoscopic approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with permanent ostomy and 1 years of life expectancy
* Signed informed consent

Exclusion Criteria:

* Allergy to the compounds of the mesh
* Rejection of the patient
* Rejection of the surgeon
* Field of emergency
* Life expectancy < 1 year
* Prior meshes in the surgical site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
If a prophylactic mesh placed through a laparoscopic approach prevents the development of a parastomal hernia when a permanent ostomy is done | 24 to 36 months after surgery

SECONDARY OUTCOMES:
Measuring the quality of life using the SF-36 | Preoperative and at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Valldhebron Research Institute, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Serra-Aracil X, Bombardo-Junca J, Moreno-Matias J, Darnell A, Mora-Lopez L, Alcantara-Moral M, Ayguavives-Garnica I, Navarro-Soto S. Randomized, controlled, prospective trial of the use of a mesh to prevent parastomal hernia. Ann Surg. 2009 Apr;249(4):583-7. doi: 10.1097/SLA.0b013e31819ec809. PMID 19300232
- [Background] Lopez-Cano M, Lozoya-Trujillo R, Espin-Basany E. Prosthetic mesh in parastomal hernia prevention. Laparoscopic approach. Dis Colon Rectum. 2009 May;52(5):1006-7. doi: 10.1007/DCR.0b013e31819a6a58. PMID 19502871
- [Derived] Lopez-Cano M, Lozoya-Trujillo R, Quiroga S, Sanchez JL, Vallribera F, Marti M, Jimenez LM, Armengol-Carrasco M, Espin E. Use of a prosthetic mesh to prevent parastomal hernia during laparoscopic abdominoperineal resection: a randomized controlled trial. Hernia. 2012 Dec;16(6):661-7. doi: 10.1007/s10029-012-0952-z. Epub 2012 Jul 11. PMID 22782367